CLINICAL TRIAL: NCT04661605
Title: Visualization Engineering Platform for Pulse Diagnosis of Traditional Chinese Medicine-The Research of Similar Moiré Feature Analyzing Approach Based on Recurrent Neural Network to Process the Measured Slip Pulse Wave-Images With Chun, Guan and Chy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMUH109-REC2-159
Record Dates: First submitted 2020-12-04; First posted 2020-12-10 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Slippery Pulse
Keywords: Artificial intelligence; Recurrent Neural Network; Wrist artery pulse diagnosis instrument; TCM pulse diagnosis; Feature extraction
MeSH Terms: interventions — Recurrent Neural Networks

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Recurrent Neural Network — We will propose a similar Moiré feature analyzing approach based on Recurrent Neural Network to process the measured Slip Pulse wave-images with 'Chun', 'Guan' and 'Chy' in order to prepare this visualization engineering platform.

SUMMARY:
The diagnoses processes of Traditional Chinese Medicine (TCM) focus on the following four main types of diagnoses methods consisting of inspection, olfaction, inquiry, and palpation. The most important one is palpation also called pulse diagnosis which is to measure wrist artery pulse by TCM doctor's fingers to detect patient's health state. The pulse diagnosis has three parts, namely 'Chun', 'Guan' and 'Chy', with the location. Wrist measurements correspond to different parts of the body's organs. However, the pulse information is analyzed by TCM doctor's pulse diagnoses process, which is picked only a single waveform from a long-term pulse measured process and often discarded the other waveforms contained in the same information, e.g. Slip Pulse waveform. The research object of this project is to divide the TCM diagnosis patients into two groups, one is the Slip pulse group and the other is a Flat Pulse group, in which the cases are collected at least 50 cases for the first gruop and 30 cases for the second group, individually. The purpose of this project will integrate the TCM doctor's experiences and standardize them in order to construct an effective Slip pulse diagnosis system based on visualization engineering platform. It could refine Slip pulse diagnoses processes and reduce their diagnoses loading by using the proposed approach during this project. Therefore, we will propose a similar Moiré feature analyzing approach based on Recurrent Neural Network to process the measured Slip Pulse wave-images with 'Chun', 'Guan' and 'Chy' in order to prepare this visualization engineering platform. We will measure the waveform images of the three parts of the wrist as 'Chun', 'Guan' and 'Chy' with the moiré feature technology proposed in this project. It mainly extracts the moiré features such as pulse image from numerous measurement 'Chun', 'Guan' and 'Chy' signals, and further analyzes and summarizes them with AI technology. We could extract the pulse characteristics of Slip pulse automatically from the many measurement signals and enhance the automatic judging ability of the current pulse instrument to the Slip pulse waveform. Provide important pulse information to the TCM doctors as an important reference for precision clinical diagnoses.

ELIGIBILITY:
Inclusion Criteria:

1. Already sign test consent permit.
2. More than 20-year-old.

Exclusion Criteria:

1. There is a wound or inflammation at the wrist skin measurement.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Outpatient.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Slippery Pulse | 30 minutes in duration
  The purpose of this project will integrate the TCM doctor's experiences and standardize them in order to construct an effective Slippery Pulse diagnosis system.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, North District, Taiwan